CLINICAL TRIAL: NCT01721954
Title: Assessment of Overall Survival of FOLFOX6m Plus SIR-Spheres Microspheres Versus FOLFOX6m Alone as First-line Treatment in Patients With Non-resectable Liver Metastases From Primary Colorectal Carcinoma in a Randomised Clinical Study
Brief Title: FOLFOX6m Plus SIR-Spheres Microspheres vs FOLFOX6m Alone in Patients With Liver Mets From Primary Colorectal Cancer
Acronym: FOXFIREGlobal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STX0112
Record Dates: First submitted 2012-10-26; First posted 2012-11-06 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Colorectal Cancer Metastatic
Keywords: colon; rectum; metastatic colorectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Active Comparator): Systemic chemotherapy with FOLFOX6m plus or minus bevacizumab repeated every two weeks until evidence of treatment failure.
  Interventions: Drug: FOLFOX6m
- Experimental Arm (Experimental): Systemic chemotherapy with FOLFOX6m plus or minus bevacizumab plus SIR-Spheres microspheres.
  Interventions: Drug: FOLFOX6m; Device: SIR-Spheres microspheres

INTERVENTIONS:
Drug: FOLFOX6m
Device: SIR-Spheres microspheres
  Arms: Experimental Arm

SUMMARY:
This study is a randomized, multi-center study that will compare the efficacy and safety of selective internal radiation therapy (SIRT) using SIR-Spheres microspheres plus a standard chemotherapy regimen of FOLFOX6m versus FOLFOX6m alone as first-line therapy in patients with non-resectable liver metastases from primary colorectal carcinoma.

Treatment with the biologic agent bevacizumab, if part of the standard of care at participating institutions, is allowed within this study at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Willing and able to provide written informed consent
* Unequivocal and measurable CT evidence of liver metastases which are not treatable by surgical resection or local ablation
* Limited extra-hepatic metastases in the lung and/or lymph nodes are permitted (Lung: 5 lesions total, < 1 cm, or 1 single lesion of up to 1.7 cm; Lymph nodules in one single anatomic area (pelvis, abdomen or chest): any number, < 2 cm)
* All imaging evidence used as part of the screening process must be within 28 days
* Suitable for either treatment regimen
* WHO performance status 0-1
* Adequate hematological, renal and hepatic function
* Life expectancy of at least 3 months without any active treatment

Exclusion Criteria:

* Evidence of ascites, cirrhosis, portal hypertension, main portal or venous involvement or thrombosis as determined by clinical or radiologic assessment
* Previous radiotherapy delivered to the liver
* Non-malignant disease that would render the patient unsuitable for treatment according to the protocol
* Peripheral neuropathy > grade 2 (NCI-CTC)
* Dose-limiting toxicity associated with previous adjuvant 5-FU or oxaliplatin chemotherapy
* Prior non-adjuvant chemotherapy for any malignancy. Adjuvant chemotherapy for colorectal cancer is permitted provided that it was completed more than 6 months before entry into the study
* Pregnant or breast feeding
* Concurrent or prior history of cancer other than adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix
* Allergy to contrast media that would preclude angiography of the hepatic arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (83):
- United States (18):
  - City of Hope, Duarte, California
  - Orlando Health, Orlando, Florida
  - Memorial Healthcare, Pembroke Pines, Florida
  - University of Illinois Chicago, Chicago, Illinois
  - Adventist Midwest Health, Hinsdale, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Roswell Park Cancer Center, Buffalo, New York
  - Lenox Hill Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Spartanburg Regional Healthcare / Gibbs Cancer Center, Spartanburg, South Carolina
  - Methodist Hospital Dallas, Dallas, Texas
  - St. Mark's Hospital, Salt Lake City, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (17):
  - Border Medical Oncology Research Unit, Albury, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Royal Brisbane Hospital, Herston, Queensland
  - Gold Coast Health Services District, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre, Bentleigh East, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Western Hospital, Footscray, Victoria
  - Peninsula Oncology Centre, Frankston, Victoria
  - South Eastern Hospital, Noble Park, Victoria
  - Maroondah Hospital, Ringwood East, Victoria
  - St. John of God Murdoch Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (6):
  - OL Vrouw Ziekenhuis, Aalst
  - Institut Jules Bordet, Brussels
  - University of Antwerp, Edegem
  - Universiteits Ziekenhuis Gent - Dienst Digestieve Oncologie, Ghent
  - AZ Maria Middelaress, Ghent
  - CHU Sart Tilman, Liège
- France (8):
  - CHU Amiens, Amiens
  - Centre Hospitalier General de Longjumeau, Clichy
  - Hopital Beaujon, Clichy
  - Hopital Albert Michallon - Grenoble, Grenoble
  - Hopital Europeen Georges Pompidou, Paris
  - CHU de Bordeaux - Hopital Saint Andre, Pessac
  - CHU de Poitiers, Pole regional de cancerologie, Poitiers
  - Centre Eugene Marquis, Rennes
- Germany (10):
  - Vivantes Klinikum Neukolln Klinik fur Innere Medizin - Hamatologie und Onkologie, Berlin
  - SLK-Kliniken Heilbronn GmbH, Klinik fur Radiologie, Heilbronn
  - Stadtisches Klinikum Karlsruheg GMBH Klinik fur Nuklearmedizin, Karlsruhe
  - Schwerpunktpraxix fur Hamatologie und Onkologie, Magdeburg
  - Universitaetsklinikum Magdeburg, Klinik fur Radiologie und Nuklearmedizin, Magdeburg
  - Klinikum Magdeburg GmbH, Klinik fur Allgemein und Viszeralchirurgie, Magdeburg
  - Universitatsklinikum Marburg Klinik fur Hamatologie, Onkologie und Immunologie, Marburg
  - Klinikum der Universitat Munchen, Munich
  - Klinikum rechts der Isar der TU Munchen Medizinische Klinik II, München
  - St. Franziskus Hospital Muenster, Münster
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare-Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - TA Sourasky Medical Center, Oncology Department 6, Tel Aviv
  - Sheba Medical Center - Governmental Hospital - Oncology Division, Tel Litwinsky
- Italy (5):
  - Ospedale Regionale U. Parini, Aosta
  - Dipartimento di Oncologia, Ospendali Riuniti di Bergamo, Bergamo
  - A.O.U. die Bologna, Bologna
  - Ufficio Sperimentale Cliniche, Oncologia Medica di Carle, Ospendale Santa Croce e Carle di Cuneo, Cuneo
  - U.O. Oncologia Medica II, Nuovo Ospendale Santa Chiara, Azienda Ospendaliero Universitaria Pisana, Presidio Ospendaliero di Cisanello, Pisa
- New Zealand (4):
  - Wellington Hospital, Newtown, Wellington Region
  - Dunedin Hospital, Dunedin
  - Auckland University, Grafton
  - Regional Cancer Treatment Service, Palmerston North
- Instituto Portugues de Oncologia do Porto Francisco Gentil, E.P.E., Porto, Portugal
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
- Spain (3):
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Complejo Hospitalario de Navarra, Pamplona
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Hazel GA, Heinemann V, Sharma NK, Findlay MP, Ricke J, Peeters M, Perez D, Robinson BA, Strickland AH, Ferguson T, Rodriguez J, Kroning H, Wolf I, Ganju V, Walpole E, Boucher E, Tichler T, Shacham-Shmueli E, Powell A, Eliadis P, Isaacs R, Price D, Moeslein F, Taieb J, Bower G, Gebski V, Van Buskirk M, Cade DN, Thurston K, Gibbs P. SIRFLOX: Randomized Phase III Trial Comparing First-Line mFOLFOX6 (Plus or Minus Bevacizumab) Versus mFOLFOX6 (Plus or Minus Bevacizumab) Plus Selective Internal Radiation Therapy in Patients With Metastatic Colorectal Cancer. J Clin Oncol. 2016 May 20;34(15):1723-31. doi: 10.1200/JCO.2015.66.1181. Epub 2016 Feb 22. PMID 26903575
- [Derived] Wolstenholme J, Fusco F, Gray AM, Moschandreas J, Virdee PS, Love S, Van Hazel G, Gibbs P, Wasan HS, Sharma RA. Quality of life in the FOXFIRE, SIRFLOX and FOXFIRE-global randomised trials of selective internal radiotherapy for metastatic colorectal cancer. Int J Cancer. 2020 Aug 15;147(4):1078-1085. doi: 10.1002/ijc.32828. Epub 2020 Jan 9. PMID 31840815
- [Derived] Wasan HS, Gibbs P, Sharma NK, Taieb J, Heinemann V, Ricke J, Peeters M, Findlay M, Weaver A, Mills J, Wilson C, Adams R, Francis A, Moschandreas J, Virdee PS, Dutton P, Love S, Gebski V, Gray A; FOXFIRE trial investigators; SIRFLOX trial investigators; FOXFIRE-Global trial investigators; van Hazel G, Sharma RA. First-line selective internal radiotherapy plus chemotherapy versus chemotherapy alone in patients with liver metastases from colorectal cancer (FOXFIRE, SIRFLOX, and FOXFIRE-Global): a combined analysis of three multicentre, randomised, phase 3 trials. Lancet Oncol. 2017 Sep;18(9):1159-1171. doi: 10.1016/S1470-2045(17)30457-6. Epub 2017 Aug 3. PMID 28781171
- [Derived] Virdee PS, Moschandreas J, Gebski V, Love SB, Francis EA, Wasan HS, van Hazel G, Gibbs P, Sharma RA. Protocol for Combined Analysis of FOXFIRE, SIRFLOX, and FOXFIRE-Global Randomized Phase III Trials of Chemotherapy +/- Selective Internal Radiation Therapy as First-Line Treatment for Patients With Metastatic Colorectal Cancer. JMIR Res Protoc. 2017 Mar 28;6(3):e43. doi: 10.2196/resprot.7201. PMID 28351831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 01May2013&24Dec2014,209 patients were screened&randomised from 87centres in Australia, Belgium,France, Germany, Israel, Italy, Korea, New Zealand, Portugal, Singapore, Spain,Taiwan &the US. 209 patients randomized in the Intent to treat (ITT) population. 5 patients who did not receive study medication were not included in safety population.
Groups:
- mFOLFOX6 Plus SIRT: Systemic chemotherapy with FOLFOX6m plus or minus bevacizumab plus SIR-Spheres microspheres.
  FOLFOX6m
  SIR-Spheres microspheres
- mFOLFOX6 Alone: Systemic chemotherapy with FOLFOX6m plus or minus bevacizumab repeated every two weeks until evidence of treatment failure.
  FOLFOX6m
Period: Overall Study
Arm/Group | mFOLFOX6 Plus SIRT | mFOLFOX6 Alone
Started | 105 | 104
Completed | 35 | 35
Not Completed | 70 | 69
Not completed — Death | 58 | 64
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mFOLFOX6 Plus SIRT | mFOLFOX6 Alone | Total
Number analyzed (Participants) | 105 | 104 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (11.28) | 62.4 (10.06) | 62.5 (10.66)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: Below 65 years | 60 | 57 | 117
  Age, Categorical: Greater than or equal to 65 years | 45 | 47 | 92
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 44 | 85
  Male | 64 | 60 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 88 | 93 | 181
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8
WHO performance status [Count of Participants; unit: Participants] — (0) Able to carry out all normal activity without restriction
  (1) Restricted in physically strenuous activity but ambulatory and able to carry out light work
  Participants
    0 | 61 | 53 | 114
    1 | 44 | 50 | 94
    Unknown | 0 | 1 | 1
Extra-hepatic Disease [Number; unit: participants]
  Yes | 32 | 27 | 59
  No | 73 | 77 | 150
Liver Involvement % [Number; unit: participants]
  <=25% | 74 | 74 | 148
  >25% | 31 | 30 | 61
Tumor volume [Mean (Standard Deviation); unit: percentage of liver] | 18.5 (17.77) | 17.9 (16.18) | 18.2 (16.96)
ITT bevacizumab [Count of Participants; unit: Participants]
  Yes | 87 | 87 | 174
  No | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS defined as the time interval between the date of randomization and the date of death from any cause.
Time Frame: From date of randomization until the date of death from any cause assessed up 3 yrs 8 months
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | mFOLFOX6 Plus SIRT | mFOLFOX6 Alone
Number analyzed (Participants) | 105 | 104
months | 25.9 [23.1 to 29.0] | 25.0 [22.1 to 28.5]
Statistical Analysis 1: Comparison: mFOLFOX6 Plus SIRT vs mFOLFOX6 Alone; The null hypothesis tested for the primary efficacy endpoint is overall survival (months) of SIRT/FOLFOX treatment versus FOLFOX is equal for both groups. The two-sided alternative hypothesis tested with 95% confidence is OS time for SIRT/FOLFOX treatment lower to that of FOLFOX; Test type: Superiority; p = 0.43, Log Rank; Hazard Ratio (HR) = 0.93

2. Secondary Outcome: Progression-free Survival
Description: PFS defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as an increase in the sum of the longest diameters of ≥ 20% and an absolute increase in the sum of the longest diameters of ≥ 5 mm, or the appearance of a new lesion.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years 8 months.
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | mFOLFOX6 Plus SIRT | mFOLFOX6 Alone
Number analyzed (Participants) | 105 | 104
months | 11.8 [10.3 to 14.5] | 11.2 [9.4 to 12.6]
Statistical Analysis 1: Comparison: mFOLFOX6 Plus SIRT vs mFOLFOX6 Alone; A sample size of at least 209 patients for the SIRFLOX study was estimated to be needed to detect an increase in the median PFS at any site from 9.4 months to 14.5 months with 80% power and 95% confidence. Taking into account the number of patients who might receive the alternative treatment or lack of imaging data, the sample size was increased to 209. The Null hypothesis is no difference between the treatment arms with respect to PFS; Test type: Superiority; p < 0.05, Log Rank; Hazard Ratio (HR) = 0.75

ADVERSE EVENTS:
Time Frame: From consent until 28 days post last dose of protocol chemotherapy, an average of 3 years 8 months.
Description: Adverse Events monitored for all participants who were randomized and received at least 1 cycle of study treatment.
  Of the 105 in 'mFOLFOX6 Plus SIRT' arm, 3 did not get any treatment,10 received mFOLFOX6 without SIRT. Hence safety population in this arm comprises 92 participants.
  The 'mFOLFOX6 alone' arm comprised 104 participants, 2 did not receive any treatment and safety population in this arm comprises 112 participants including the 10 participants that received mFOLFOX6 without SIRT.
Arm/Group | mFOLFOX6 Plus SIRT | mFOLFOX6 Alone
All-Cause Mortality (participants affected / at risk) | 58/92 | 64/112
Serious Adverse Events (participants affected / at risk) | 47/92 | 47/112
Other Adverse Events (participants affected / at risk) | 92/92 | 111/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 Plus SIRT (N=92) | mFOLFOX6 Alone (N=112)
Febrile Neutropenia (Blood and lymphatic system disorders) | 10 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Arteriospasm Coronary (Cardiac disorders) | 1 | 1
Cardiac Failure (Cardiac disorders) | 0 | 1
Cardiotoxicity (Cardiac disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 9 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Duodenal Perforation (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Neutropenic Colitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Varices Oesophageal (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
General Physical Health Deterioration (General disorders) | 2 | 2
Malaise (General disorders) | 1 | 1
Mucosal Inflammation (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 2 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Portal Hypertension (Hepatobiliary disorders) | 0 | 1
Abdominal Sepsis (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 1
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 1 | 1
Device Related Sepsis (Infections and infestations) | 0 | 1
Enteritis Infectious (Infections and infestations) | 0 | 1
Enterococcal Sepsis (Infections and infestations) | 1 | 0
Escherichia Sepsis (Infections and infestations) | 2 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Infusion Site Cellulitis (Infections and infestations) | 1 | 0
Infusion Site Infection (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1
Lung Abscess (Infections and infestations) | 0 | 1
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Pelvic Abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Peritonitis Bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 3
Pseudomonal Bacteraemia (Infections and infestations) | 1 | 0
Rectal Abscess (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 2
Skin Bacterial Infection (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 2
Arterial Injury (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 | 2
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Intestinal Anastomosis Complication (Injury, poisoning and procedural complications) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Diabetic Complication (Metabolism and nutrition disorders) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Encephalopathy (Nervous system disorders) | 2 | 0
Mental Impairment (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Acute Psychosis (Psychiatric disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 2
Delirium (Psychiatric disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Renal Injury (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Artery Dissection (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Jugular Vein Thrombosis (Vascular disorders) | 0 | 1
Orthostatic Hypotensio (Vascular disorders) | 1 | 1
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 0
Vena Cava Thrombosis (Vascular disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 Plus SIRT (N=92) | mFOLFOX6 Alone (N=112)
Neutropenia (Blood and lymphatic system disorders) | 43 | 46
Thrombocytopenia (Blood and lymphatic system disorders) | 39 | 11
Anaemia (Blood and lymphatic system disorders) | 21 | 15
Leukopenia (Blood and lymphatic system disorders) | 13 | 10
Lymphopenia (Blood and lymphatic system disorders) | 6 | 1
Lacrimation Increased (Eye disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 46 | 55
Diarrhoea (Gastrointestinal disorders) | 35 | 59
Constipation (Gastrointestinal disorders) | 39 | 45
Abdominal Pain (Gastrointestinal disorders) | 33 | 24
Vomiting (Gastrointestinal disorders) | 24 | 33
Stomatitis (Gastrointestinal disorders) | 21 | 29
Abdominal Pain Upper (Gastrointestinal disorders) | 20 | 12
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 7 | 14
Mouth Ulceration (Gastrointestinal disorders) | 4 | 14
Abdominal Distension (Gastrointestinal disorders) | 9 | 7
Rectal Haemorrhage (Gastrointestinal disorders) | 7 | 7
Dry Mouth (Gastrointestinal disorders) | 3 | 9
Ascites (Gastrointestinal disorders) | 9 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 5
Gastritis (Gastrointestinal disorders) | 5 | 1
Fatigue (General disorders) | 48 | 49
Mucosal Inflammation (General disorders) | 12 | 23
Asthenia (General disorders) | 15 | 18
Pyrexia (General disorders) | 17 | 16
Oedema Peripheral (General disorders) | 13 | 6
Pain (General disorders) | 3 | 8
Chest Pain (General disorders) | 1 | 8
Urinary Tract Infection (Infections and infestations) | 9 | 10
Upper Respiratory Tract Infection (Infections and infestations) | 10 | 8
Nasopharyngitis (Infections and infestations) | 2 | 8
Bronchitis (Infections and infestations) | 1 | 6
Contusion (Injury, poisoning and procedural complications) | 5 | 3
Fall (Injury, poisoning and procedural complications) | 5 | 2
Weight Decreased (Investigations) | 29 | 19
Neutrophil Count Decreased (Investigations) | 7 | 8
Weight Increased (Investigations) | 5 | 9
Platelet Count Decreased (Investigations) | 9 | 4
Aspartate Aminotransferase Increased (Investigations) | 9 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 6 | 5
White Blood Cell Count Decreased (Investigations) | 7 | 4
Blood Bilirubin Increased (Investigations) | 5 | 3
Alanine Aminotransferase Increased (Investigations) | 6 | 1
Blood Albumin Decreased (Investigations) | 5 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 25 | 30
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 13
Dehydration (Metabolism and nutrition disorders) | 5 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 14
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 | 12
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 13 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 8
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 7
Insomnia (Psychiatric disorders) | 16 | 15
Anxiety (Psychiatric disorders) | 8 | 12
Dysuria (Renal and urinary disorders) | 1 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 11 | 19
Rash (Skin and subcutaneous tissue disorders) | 13 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 15
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7
Hypertension (Vascular disorders) | 15 | 28
Neuropathy peripheral (Nervous system disorders) | 54 | 55
Peripheral sensory neuropathy (Nervous system disorders) | 16 | 29
Headache (Nervous system disorders) | 13 | 21
Paraesthesia (Nervous system disorders) | 15 | 19
Dysgeusia (Nervous system disorders) | 17 | 10
Dizziness (Nervous system disorders) | 8 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No